CLINICAL TRIAL: NCT00535977
Title: A Human Intervention Trial Studying Gene Expression in High-Grade Prostatic Intraepithelial Neoplasia Following Consumption of Broccoli or Peas
Brief Title: Broccoli, Peas and PIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IFR07-2004; 05/Q0101/9; 2004IFR04
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Prostatic Intraepithelial Neoplasia
Keywords: Gene expression; Prostate; Broccoli; Cancer; Men diagnosed with high-grade Prostatic Intraepithelia Neoplasia
MeSH Terms: conditions — Prostatic Intraepithelial Neoplasia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dietary intervention of ITC-enriched broccoli
  Interventions: Dietary Supplement: Broccoli
- 2 (Experimental): Dietary intervention of frozen peas
  Interventions: Dietary Supplement: Peas

INTERVENTIONS:
Dietary Supplement: Broccoli — 400g ITC-enriched broccoli per week for 12 months
  Arms: 1
Dietary Supplement: Peas — 400g frozen garden peas per week for 12 months
  Arms: 2

SUMMARY:
This is a parallel human intervention trial to determine to what extent a dietary intervention of broccoli or peas can change the expression (switching on or off) of genes in prostate tissue in men diagnosed with high-grade Prostate Intraepithelial Neoplasia (PIN).

DETAILED DESCRIPTION:
Cancer is one of the main causes of death among humans in the world. Prostate cancer affects 20,000 men in the UK alone each year. Diet is known to be a major factor that influences risk of cancer. Therefore, changes to the diet may alter cancer risk. Cruciferous vegetables, particularly broccoli, provide the diet with a substantial source of plant chemicals called glucosinolates. Previous research has indicated that glucosinolates break down to form isothiocyanates (ITCs) that can be absorbed in the body. Further research has indicated that ITCs may protect the body against the development of prostate cancer. However, the mechanisms behind this effect are not fully understood.

ITCs are thought to be powerful anti cancer agents as they can modulate the expression (switching on or off) of specific genes involved in the removal of toxic substances such as carcinogens from the body. In this study we wish to evaluate the effect of consumption of a conventionally bred cultivar of broccoli containing high levels of ITCs on gene expression in prostate tissue to gain a better understanding of its mechanism of action. Several studies suggest a further protection against cancer amongst individuals who have a deletion of certain genes.

This pilot study comprises a 12-month intervention of either 400g ITC-enriched broccoli per week of 400g garden peas in men at high risk of developing prostate cancer. Changes in gene expression of prostate biopsy tissue will be compared before and after 6 and 12 months of intervention in both dietary groups.

ELIGIBILITY:
Inclusion Criteria:

* Men with a previous diagnosis of high-grade Prostatic Intraepithelial Neoplasia
* BMI >18.5 or <35
* Aged between 30-70 years

Exclusion Criteria:

* Undergoing chemopreventive therapy
* Receiving testosterone replacement medicines
* Active infection requiring treatment
* BMI <18.5 or >35
* Diagnosed with diabetes
* Unable to give informed consent

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in RNA extracted from prostate tissue | Baseline, 6 months and 12 months

SECONDARY OUTCOMES:
Changes in levels of serum prostate specific antigen (PSA) | Baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Mithen, PhD, Principal Investigator — Institute of Food Research, Norwich

REFERENCES:
- [Background] Chiao JW, Chung FL, Kancherla R, Ahmed T, Mittelman A, Conaway CC. Sulforaphane and its metabolite mediate growth arrest and apoptosis in human prostate cancer cells. Int J Oncol. 2002 Mar;20(3):631-6. doi: 10.3892/ijo.20.3.631. PMID 11836580
- [Background] Cotton SC, Sharp L, Little J, Brockton N. Glutathione S-transferase polymorphisms and colorectal cancer: a HuGE review. Am J Epidemiol. 2000 Jan 1;151(1):7-32. doi: 10.1093/oxfordjournals.aje.a010124. PMID 10625170
- [Background] Fenwick GR, Heaney RK, Mullin WJ. Glucosinolates and their breakdown products in food and food plants. Crit Rev Food Sci Nutr. 1983;18(2):123-201. doi: 10.1080/10408398209527361. No abstract available. PMID 6337782
- [Background] Gamet-Payrastre L, Li P, Lumeau S, Cassar G, Dupont MA, Chevolleau S, Gasc N, Tulliez J, Terce F. Sulforaphane, a naturally occurring isothiocyanate, induces cell cycle arrest and apoptosis in HT29 human colon cancer cells. Cancer Res. 2000 Mar 1;60(5):1426-33. PMID 10728709
- [Background] Giovannucci E, Rimm EB, Liu Y, Stampfer MJ, Willett WC. A prospective study of cruciferous vegetables and prostate cancer. Cancer Epidemiol Biomarkers Prev. 2003 Dec;12(12):1403-9. PMID 14693729
- [Background] Hecht SS. Inhibition of carcinogenesis by isothiocyanates. Drug Metab Rev. 2000 Aug-Nov;32(3-4):395-411. doi: 10.1081/dmr-100102342. PMID 11139137
- [Background] Hintze KJ, Keck AS, Finley JW, Jeffery EH. Induction of hepatic thioredoxin reductase activity by sulforaphane, both in Hepa1c1c7 cells and in male Fisher 344 rats. J Nutr Biochem. 2003 Mar;14(3):173-179. doi: 10.1016/s0955-2863(02)00282-6. PMID 12742546
- [Background] Key TJ, Silcocks PB, Davey GK, Appleby PN, Bishop DT. A case-control study of diet and prostate cancer. Br J Cancer. 1997;76(5):678-87. doi: 10.1038/bjc.1997.445. PMID 9303371
- [Background] Mithen R, Faulkner K, Magrath R, Rose P, Williamson G, Marquez J. Development of isothiocyanate-enriched broccoli, and its enhanced ability to induce phase 2 detoxification enzymes in mammalian cells. Theor Appl Genet. 2003 Feb;106(4):727-34. doi: 10.1007/s00122-002-1123-x. Epub 2002 Oct 24. PMID 12596003
- [Background] Surh YJ. Cancer chemoprevention with dietary phytochemicals. Nat Rev Cancer. 2003 Oct;3(10):768-80. doi: 10.1038/nrc1189. PMID 14570043
- [Derived] Traka M, Gasper AV, Melchini A, Bacon JR, Needs PW, Frost V, Chantry A, Jones AM, Ortori CA, Barrett DA, Ball RY, Mills RD, Mithen RF. Broccoli consumption interacts with GSTM1 to perturb oncogenic signalling pathways in the prostate. PLoS One. 2008 Jul 2;3(7):e2568. doi: 10.1371/journal.pone.0002568. PMID 18596959